CLINICAL TRIAL: NCT04445415
Title: Diagnostic Value of New- Covid 19 Antibodies Testing Among Laboratory Healthcare Workers
Brief Title: Diagnostic Value of New COVID-19 Antibodies Testing Among Laboratory Healthcare Workers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samar Salah Eldin Abdelrahman Sultan, Resident physician, Assiut University
Other Study IDs: COVID-19 antibodies testing
Record Dates: First submitted 2020-06-18; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: COVID-19 antibodies testing — antibodies aganist COVID-19 detected in the serum of patients

SUMMARY:
COVID-19 antibodies testing among healthcare workers to evaluate the role of Covid 19Ab testing as screening method for detection of covid 19 infections among laboratory health care workers ,assess the relationship between the infection with Covid 19 and different laboratory categories/area and assessemt of efficiency personal protective equipment (PPE) in different laboratory categories/area.

DETAILED DESCRIPTION:
In December 2019, a new corona virus (CoV) emerged in China to cause an acute respiratory disease known as corona virus disease 19 (COVID-19).The virus was identified to be a betacoronavirus related to severe acute respiratory syndrome corona virus (SARS-CoV) and thus, was named SARS-CoV-2 .

New Covid-19 virus is the third known corona virus to cross the species barrier and cause severe respiratory infections in humans following SARS-CoV in 2003 and Middle East respiratory syndrome in 2012, yet with pandemic spread compared to the earlier two. In comparison, to SARS-CoV and MERS-CoV, COVID-19 virus exhibits faster human-to-human transmission.

The World Health Organization (WHO) declared COVID-19 outbreak as a world pandemic on 12th March 2020. Diagnosis of suspected cases is confirmed by molecular techniques (real-time PCR), using respiratory samples. Serology tests are easier to perform than molecular testing, but their utility may be limited by the performance and the fact that antibodies appear later during the disease course.

In the absence of a vaccine, public health authorities in several countries has shown that shutdowns can only be safely ended if a systematic "test and trace" program is put in place to control the spread of the virus which depends on the widespread availability of mass diagnostic testing.

From this point of view, detecting carriers of the virus in asymptomatic laboratory health care worker is fundamental to response efforts. It ensures the quarantine of COVID-19 patients to prevent local spread and more broadly informs national response measures.

The main route of transmission is person-to-person spread. A vulnerable cohort for infection due to frequent and close contact to COVID-19 patients are healthcare workers. To avoid patient-to-staff transmission adherence to strict hygiene standards is important. The infection with the SARS-CoV-2 usually leads to seroconversion 11-14 days after the first symptoms . However, due to asymptomatic and oligosymptomatic infections testing only symptomatic individuals can lead to a significant underestimation of the SARS-CoV-2 seroprevalence Day,.

Antibody testing is multipurpose: these serological assays are of critical importance to determine seroprevalence, previous exposure and identify highly reactive human donors for the generation of convalescent serum as therapeutic. They will support contact tracing and screening of health care workers to identify those who are already immune. How many people really got infected, in how many did the virus escape the PCR diagnosis, and for what reasons, how many patients are asymptomatic, and what is the real mortality rate in a defined population? Only with comprehensive serology testing (and well-planned epidemiological studies) will we be able to answer these questions and reduce the ubiquitous undisclosed number in the current calculations. Several investigations are already underway in a wide variety of locations worldwide

ELIGIBILITY:
Inclusion Criteria:

* • Covid 19 infected healthcare workers.

Exclusion Criteria:

* •Risky healthcare workers (diabetic, hypertensive and more than 50 years)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: the study was carried out using EPI info 2000 statistical package and based on a CDC COVID-19 Response Team report where the prevalence of COVID 19 infected health care workers (CDC, 2020) The minimum calculated sample was 250 health care worker , with confidence interval 80%.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic value of COVID-19 antibodies testing | baseline
  these serological assays are of critical importance to determine previous exposure,How many people really got infected, and for what reasons, how many patients are asymptomatic, and what is the real mortality rate in a defined population
Role of COVID -19 Antibodies testing in treatment of Patients | Baseline
  these serological assays are of critical importance to determine seroprevalence, previous exposure and identify highly reactive human donors for the generation of convalescent serum as therapeutic method for infected persons
Assement of COVID -19 prevalence among healthcare workers | Baseline
  Serological assay of COVID-19 antibodies testing will support contact tracing and screening of health care workers to identify those who are already immune. How many people really got infected, in how many did the virus escape the PCR diagnosis, and for what reasons, how many patients are asymptomatic, and what is the real mortality rate in a defined population

REFERENCES:
- [Background] Zainol Rashid Z, Othman SN, Abdul Samat MN, Ali UK, Wong KK. Diagnostic performance of COVID-19 serology assays. Malays J Pathol. 2020 Apr;42(1):13-21. PMID 32342927
- [Background] Salathe M, Althaus CL, Neher R, Stringhini S, Hodcroft E, Fellay J, Zwahlen M, Senti G, Battegay M, Wilder-Smith A, Eckerle I, Egger M, Low N. COVID-19 epidemic in Switzerland: on the importance of testing, contact tracing and isolation. Swiss Med Wkly. 2020 Mar 19;150:w20225. doi: 10.4414/smw.2020.20225. eCollection 2020 Mar 9. PMID 32191813
- [Background] Day M. Covid-19: identifying and isolating asymptomatic people helped eliminate virus in Italian village. BMJ. 2020 Mar 23;368:m1165. doi: 10.1136/bmj.m1165. No abstract available. PMID 32205334
- [Background] Long QX, Liu BZ, Deng HJ, Wu GC, Deng K, Chen YK, Liao P, Qiu JF, Lin Y, Cai XF, Wang DQ, Hu Y, Ren JH, Tang N, Xu YY, Yu LH, Mo Z, Gong F, Zhang XL, Tian WG, Hu L, Zhang XX, Xiang JL, Du HX, Liu HW, Lang CH, Luo XH, Wu SB, Cui XP, Zhou Z, Zhu MM, Wang J, Xue CJ, Li XF, Wang L, Li ZJ, Wang K, Niu CC, Yang QJ, Tang XJ, Zhang Y, Liu XM, Li JJ, Zhang DC, Zhang F, Liu P, Yuan J, Li Q, Hu JL, Chen J, Huang AL. Antibody responses to SARS-CoV-2 in patients with COVID-19. Nat Med. 2020 Jun;26(6):845-848. doi: 10.1038/s41591-020-0897-1. Epub 2020 Apr 29. PMID 32350462